CLINICAL TRIAL: NCT01442103
Title: Open, Non Comparative, Single Center Investigation Exploring the Clinical Utility of a New Silver Gel for Use on Chronic Wounds
Brief Title: Clinical Utility of a New Silver Gel for Use on Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ngel Ag 01
Record Dates: First submitted 2011-09-13; First posted 2011-09-28 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device, dressing (Experimental): Normlgel Ag is an opaque, amorphous hydrogel containing a high water content, water soluble polymer chains and an antimicrobial silver compound.
  Interventions: Device: Normlgel Ag

INTERVENTIONS:
Device: Normlgel Ag — Normlgel Ag dressing will be changed together with planned investigation visits. Dressing changes between visits will be performed at home on Day 3 or 4 of each week by subject or caregiver and documented in a dressing log.

SUMMARY:
This investigation will be conducted in the US as a single-center study to evaluate in total 10 subjects, to explore the clinical utility of a new silver gel for use on chronic wounds.

DETAILED DESCRIPTION:
Both inpatients and outpatients will be included in this study. The patients will present with chronic wounds in need of initial treatment prior to initiating standard of care (i.e. wound bed with eschar or slough), in need of treatment after debridement or with presenting inflammation along with need for treatment.Only one wound will be chosen for treatment in the study and the area should not exceed 10x10 cm and not be deeper than 6 cm. Photos of the wound will be taken at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Both genders with an age >18 years
3. Subjects with chronic wounds < 1 year chronicity that are assessed as having localized infection or inflammation (i.e. not felt to have systemic involvement) as indicated by the presence of at least 2 of the following clinical signs of infection:

   * Erythema
   * Edema
   * Warmth
   * Increased drainage
   * Foul odor
4. Subject's wounds may also present with:

   * presence of eschar or slough that needs to be treated prior to normal standard of care OR
   * A need for topical care after debridement
5. Study site to include only ONE wound to be treated

Exclusion Criteria:

1. Presence of fever with 2 or more clinical signs of infection that in the opinion of the investigator is indicative of a more systemic type infection.
2. Use of anti-microbial dressings or topical agents such as antiseptics, local antibiotics and steroids within 7 days
3. Wound > 1 year old
4. Wound > 10 cm x 10 cm (l x w)
5. Wound > 6 cm deep
6. Use of chemical/enzymatic and biological debridement within 7 days of investigation start
7. Necrotizing wounds
8. Diagnosed underlying disease(s) (e.g. HIV/AIDS, cancer and severe anaemia) judged by the investigator to be a potential interference in the treatment.
9. Subjects with poorly controlled diabetes mellitus (as judged by the investigator).
10. Subjects treated with systemic glucocorticosteroids, except subjects taking occasional doses or doses less than 10mg prednisone/day or equivalent.
11. Known allergy/hypersensitivity to any of the components of the investigation products.
12. Subjects with physical and/or mental conditions that are not expected to comply with the investigation, including subjects totally confined to bed.
13. Participation in other clinical investigation(s) within 1 month prior to Previously randomized to this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaheed Hassan, MD, Principal Investigator — Josepth M. Still Research Foundation, Augusta, Georgia, US
Locations (1):
- Joseph M. Still Research Foundation, Inc., Augusta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 15 September 2011 - 01 May 2012. The study was conducted at the Advanced Burn and Wound Clinic at the Joseph M. Still Burn Center in Augusta, Georgia.
Pre-assignment Details: PreAssignment details:
  There was not wash-out or run-in phase included in the study. Subjects were expected to have at least 2 signs of local irritation or inflammation but no active or systemic infection at the time of consent.
Groups:
- Silver Gel, Chronic Wounds: The patients will present with chronic wounds in need of initial treatment prior to initiating standard of care (i.e. wound bed with eschar or slough), in need of treatment after debridement or with presenting inflammation along with need for treatment.Only one wound will be chosen for treatment in the study and the area should not exceed 10x10 cm and not be deeper than 6 cm. Photos of the wound will be taken at each visit.
Period: Overall Study
Arm/Group | Silver Gel, Chronic Wounds
Started | 10
Completed | 8
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Silver Gel, Chronic Wounds: Open, non-comparative, single-centre investigation exploring the clinical utility of a new silver gel for use on chronic wounds.
Arm/Group | Silver Gel, Chronic Wounds
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Signs and Symptoms of Local Wound Infection/Inflammation.
Description: Signs and symptoms of local wound infection/inflammation will be assessed by visual infection assessment (including body temperature) and wound status.
Time Frame: 4 weeks
Population: Popul for the asses.of safety was incld all subjs that received at least one device and that provided data after baseline. Prim.analys:ITT, popul incld all subjs that provid.data for the prim endpoint Parameters were summ for the ITT popul using apt sum. statistics. Data described in a descriptive manner only. Efficacy endpoints were sum.by visit.
Measure: Number; unit: participants
Groups:
- Device Common Dressing: Normlgel® Ag is an opaque, amorphous hyrdrogel containing a high (>80%) water content and water soluble polymer chains.
Arm/Group | Device Common Dressing
Number analyzed (Participants) | 10
participants | 8

2. Secondary Outcome: Infection Assessment
Description: Erythema, edema, warmth, increased drainage, foul odor and fever will be assessed at each visit.
Time Frame: 4 weekks
Reporting Status: Not Posted

3. Secondary Outcome: Pain Upon Application of Investigational Product.
Description: VAS pain scale will be used to measuring pain at each dressing change.
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Device Common Dressing: Normal Ag is an opaque, amorphous hydrogel containing a high watersoluble polymer chains and an antimicrobial silver compund
Arm/Group | Device Common Dressing
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Small study population, 2 patients lost to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No